CLINICAL TRIAL: NCT01362062
Title: A Study to Observe the Safety, Tolerability and Efficacy of Tocilizumab in Patients With Moderate to Severe Active Rheumatoid Arthritis Who Have an Inadequate Response to Current Non-biologic DMARD and/or Anti TNF Therapy.
Brief Title: Study to Evaluate the Safety, Tolerability and Efficacy of Tocilizumab in Participants With Rheumatoid Arthritis (RA) Who Have an Inadequate Response to Non-Biologic Disease Modifying Anti-rheumatic Drugs (DMARDs) and/or Anti-tumor Necrosis Factor (Anti-TNF) Therapy
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML22835
Record Dates: First submitted 2011-05-26; First posted 2011-05-27 (Estimated); Results first posted 2016-04-04 (Estimated); Last update posted 2017-08-02 (Actual); Status verified 2017-06

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- RA Cohort: Participants with active RA who had an inadequate clinical response to current non-biologic disease modifying anti-rheumatoid drug (DMARD) and/or anti-tumor necrosis factor (anti-TNF) therapy being treated with tocilizumab according to the routine clinical practice and in line with prescribing information will be observed for a total duration of 12 months.
  Interventions: Drug: Tocilizumab

INTERVENTIONS:
Drug: Tocilizumab
  Other Names: Actemra

SUMMARY:
This observational study will evaluate the safety, tolerability and efficacy of tocilizumab in participants with moderate to severe RA who have an inadequate response to current non-biologic DMARD and/or anti-TNF therapy. Data will be collected from each participant during tocilizumab therapy and on follow-up for a total of 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe active RA with an inadequate response to existing therapies (DMARDs and/or anti-TNFs)
* Considered eligible for tocilizumab therapy by the treating physician as per routine clinical practice

Exclusion Criteria:

* Pregnant or breastfeeding females
* Immunization with live/attenuated vaccine within 4 weeks prior to baseline
* Participants with clinically significant raised liver enzyme, abnormal lipid profile, platelet count, hemoglobin, white blood cell and neutrophil count
* History of severe allergic or anaphylactic reactions to human, humanized or murine monoclonal antibodies
* Participants with active tuberculosis (TB). Participants with latent TB should be treated with standard anti-mycobacterial therapy before initiating tocilizumab and have a negative chest x ray for active TB at enrolment
* History of diverticulitis, chronic ulcerative lower GI disease such as Crohn's disease, ulcerative colitis or other symptomatic lower GI conditions that might predispose to perforations then the benefit risk ratio should be considered by treating physician
* Know active current or history of recurrent bacterial, viral, fungal, mycobacterial or other infection
* History of or currently active primary or secondary immunodeficiency or known human immunodeficiency virus (HIV) positive status
* Any other condition which puts the participant to undue risk for tocilizumab therapy as per local prescribing information or Investigator's judgement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Rheumatoid arthritis patients with inadequate response to DMARD and/or anti-TNF therapy
Sampling Method: Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2010-10-26 (Actual); Primary Completion 2015-01-01 (Actual); Study Completion 2015-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (7):
- India (7):
  - Sir Gangaram Hospital, New Delhi, National Capital Territory of Delhi
  - Healing Touch City Clinic, Chandigarh
  - Excel Center, Guwahati
  - Arthritis Superspeciality Centre, Hubli
  - Centre for Rheumatic Diseases - Mumbai, Mumbai
  - Jivdaya Clinic, Mumbai
  - Fortis Hospital, Noida

RESULTS

PARTICIPANT FLOW:
Groups:
- RA Cohort (Prospective): Participants with active RA who had an inadequate clinical response to current non-biologic disease modifying anti-rheumatoid drug (DMARD) and/or anti-tumor necrosis factor (anti-TNF) therapy being treated with tocilizumab according to the routine clinical practice and in line with prescribing information were observed prospectively for a total duration of 12 months.
- RA Cohort (Retrospective): Participants with active RA who had an inadequate clinical response to current non-biologic DMARD and/or anti-TNF therapy being treated with tocilizumab according to the routine clinical practice and in line with prescribing information were observed retrospectively for a total duration of 12 months.
Period: Overall Study
Arm/Group | RA Cohort (Prospective) | RA Cohort (Retrospective)
Started | 48 | 62
Completed | 22 | 62
Not Completed | 26 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 11 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Non-compliant participant | 2 | 0
Not completed — Detected with Spondylo-arthritis | 1 | 0
Not completed — Had significant improvement | 9 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants who were considered evaluable for analysis.
Groups:
- RA Cohort (Prospective): Participants with active RA who had an inadequate clinical response to current non-biologic DMARD and/or anti-TNF therapy being treated with tocilizumab according to the routine clinical practice and in line with prescribing information were observed prospectively for a total duration of 12 months.
- Total: Total of all reporting groups
Arm/Group | RA Cohort (Prospective) | RA Cohort (Retrospective) | Total
Number analyzed (Participants) | 48 | 62 | 110
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.19 (10.44) | 50.39 (12.56) | 50.74 (11.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 54 | 94
  Male | 8 | 8 | 16

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Events (AEs) or Serious AEs (SAEs)
Description: An AE is any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not considered related to the medicinal product. An AE is considered as an SAE if it fulfills one of the following criteria: a) fatal or life-threatening, b) requires in-patient hospitalization or prolongation of existing hospitalization, c) results in a persistent or significant disability, d) results in a congenital abnormality/birth defect, e) is medically significant. AEs included serious as well as non-serious AEs.
Time Frame: Up to 12 months
Population: Safety analysis population: Included all participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Groups:
- RA Cohort (Prospective + Retrospective): Participants with active RA who had an inadequate clinical response to current non-biologic DMARD and/or anti-TNF therapy being treated with tocilizumab according to the routine clinical practice and in line with prescribing information were observed prospectively or retrospectively for a total duration of 12 months.
Arm/Group | RA Cohort (Prospective + Retrospective)
Number analyzed (Participants) | 110
percentage of participants
  AEs | 31.8
  SAEs | 7.2

2. Secondary Outcome: Percentage of Participants Achieving a Clinically Meaningful Improvement in Disease Activity Score 28 (DAS28) (Reduction of At Least 1.2 Units) at Every Visit
Description: DAS28 was calculated from the tender joint count (TJC) of 28 joints, swollen joint count (SJC) of 28 joints, erythrocyte sedimentation rate (ESR) (in millimeters [mm]/hour), and the participant's global assessment of disease activity (100 mm visual analog scale [VAS]: 0 mm=no disease activity to 100 mm=maximum disease activity). The formula for calculating DAS28 score using ESR value is: 0.56*square root (√) of TJC + 0.28*√(SJC) + 0.70*log natural (ESR) + 0.014*global assessment of disease activity (100 mm VAS). The DAS28 scale ranges from 0 to 10, where higher scores represent higher disease activity. A reduction of at least 1.2 units of DAS28 score from previous visit is considered as clinically meaningful improvement.
Time Frame: Visit 3 (Week 4), Visit 4 (Week 8), Visit 5 (Week 12), Visit 6 (Week 16), Visit 7 (Week 20), Visit 8 (Week 24), Visit 9 (Week 28), Visit 10 (Week 32), Visit 11 (Week 36), Visit 12 (Week 40), Visit 13 (Week 44)
Population: Efficacy analysis population included participants who were observed prospectively in this study. Number of participants analyzed = number of participants evaluable for this outcome and n = number of participants evaluable at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | RA Cohort (Prospective)
Number analyzed (Participants) | 43
percentage of participants
  Visit 3 (n=38) | 55.3
  Visit 4 (n=37) | 73.0
  Visit 5 (n=37) | 81.1
  Visit 6 (n=36) | 80.6
  Visit 7 (n=39) | 84.6
  Visit 8 (n=21) | 90.5
  Visit 9 (n=20) | 85.0
  Visit 10 (n=18) | 88.9
  Visit 11 (n=23) | 87.0
  Visit 12 (n=20) | 95.0
  Visit 13 (n=17) | 94.1
  Overall (n=43) | 97.7

3. Secondary Outcome: Time Required to Achieve Clinically Meaningful Improvement in DAS28 (Reduction of At Least 1.2 Units)
Description: DAS28 was calculated from the TJC of 28 joints, SJC of 28 joints, ESR (in mm/hour), and the participant's global assessment of disease activity (100 mm VAS: 0 mm=no disease activity to 100 mm=maximum disease activity). The formula for calculating DAS28 score using ESR value is: 0.56*√(TJC) + 0.28*√(SJC) + 0.70*log natural (ESR) + 0.014*global assessment of disease activity (100 mm VAS). The DAS28 scale ranges from 0 to 10, where higher scores represent higher disease activity. A reduction of at least 1.2 units of DAS28 score from previous visit is considered as clinically meaningful improvement. Time taken to achieve clinically meaningful improvement in DAS28 was reported.
Time Frame: Up to 12 months
Population: Efficacy analysis population. Number of participants analyzed = number of participants evaluable for this outcome.
Measure: Mean (Full Range); unit: days
Arm/Group | RA Cohort (Prospective)
Number analyzed (Participants) | 43
days | 60 [28 to 252]

4. Secondary Outcome: Percentage of Participants Achieving Low Disease Activity (DAS28 Less Than [<] 3.2 Units) at Every Visit
Description: DAS28 was calculated from the TJC of 28 joints, SJC of 28 joints, ESR (in mm/hour), and the participant's global assessment of disease activity (100 mm VAS: 0 mm=no disease activity to 100 mm=maximum disease activity). The formula for calculating DAS28 score using ESR value is: 0.56*√(TJC) + 0.28*√(SJC) + 0.70*log natural (ESR) + 0.014*global assessment of disease activity (100 mm VAS). The DAS28 scale ranges from 0 to 10, where higher scores represent higher disease activity. Low Disease Activity is defined as DAS28 value of <3.2 Units at the time of assessment.
Time Frame: as for outcome 2
Population: Efficacy analysis population. Number of participants analyzed = number of participants evaluable for this outcome and n = number of participants evaluable at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | RA Cohort (Prospective)
Number analyzed (Participants) | 43
percentage of participants
  Visit 3 (n=38) | 15.8
  Visit 4 (n=37) | 27.0
  Visit 5 (n=37) | 29.7
  Visit 6 (n=36) | 44.4
  Visit 7 (n=39) | 46.2
  Visit 8 (n=21) | 42.9
  Visit 9 (n=20) | 45.0
  Visit 10 (n=18) | 50.0
  Visit 11 (n=23) | 60.9
  Visit 12 (n=20) | 70.0
  Visit 13 (n=17) | 64.7
  Overall (n=43) | 74.4

5. Secondary Outcome: Time Required to Achieve Low Disease Activity (DAS28 <3.2 Units)
Description: DAS28 was calculated from the TJC of 28 joints, SJC of 28 joints, ESR (in mm/hour), and the participant's global assessment of disease activity (100 mm VAS: 0 mm=no disease activity to 100 mm=maximum disease activity). The formula for calculating DAS28 score using ESR value is: 0.56*√(TJC) + 0.28*√(SJC) + 0.70*log natural (ESR) + 0.014*global assessment of disease activity (100 mm VAS). The DAS28 scale ranges from 0 to 10, where higher scores represent higher disease activity. Low disease activity is defined as decrease in DAS28 to a value <3.2 Units at the time of assessment. Time taken to achieve low disease activity was reported.
Time Frame: Up to 12 months
Population: Efficacy analysis population. Number of participants analyzed = number of participants evaluable for this outcome.
Measure: Mean (Full Range); unit: days
Arm/Group | RA Cohort (Prospective)
Number analyzed (Participants) | 43
days | 117.25 [28 to 252]

6. Secondary Outcome: Percentage of Participants Achieving Remission (DAS28 <2.6 Units) at Every Visit
Description: DAS28 was calculated from the TJC of 28 joints, SJC of 28 joints, ESR (in mm/hour), and the participant's global assessment of disease activity (100 mm VAS: 0 mm=no disease activity to 100 mm=maximum disease activity). The formula for calculating DAS28 score using ESR value is: 0.56*√(TJC) + 0.28*√(SJC) + 0.70*log natural (ESR) + 0.014*global assessment of disease activity (100 mm VAS). Remission is defined as DAS28 value of <2.6 units at the time of assessment.
Time Frame: as for outcome 2
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | RA Cohort (Prospective)
Number analyzed (Participants) | 43
percentage of participants
  Visit 3 (n=38) | 5.3
  Visit 4 (n=37) | 10.8
  Visit 5 (n=37) | 16.2
  Visit 6 (n=36) | 30.6
  Visit 7 (n=39) | 35.9
  Visit 8 (n=21) | 28.6
  Visit 9 (n=20) | 35.0
  Visit 10 (n=18) | 38.9
  Visit 11 (n=23) | 52.2
  Visit 12 (n=20) | 55.0
  Visit 13 (n=17) | 58.8
  Overall (n=43) | 60.5

7. Secondary Outcome: Time Taken to Achieve Remission (DAS28 <2.6 Units)
Description: DAS28 was calculated from the TJC of 28 joints, SJC of 28 joints, ESR (in mm/hour), and the participant's global assessment of disease activity (100 mm VAS: 0 mm=no disease activity to 100 mm=maximum disease activity). The formula for calculating DAS28 score using ESR value is: 0.56*√(TJC) + 0.28*√(SJC) + 0.70*log natural (ESR) + 0.014*global assessment of disease activity (100 mm VAS). Remission is defined as DAS28 value of <2.6 units at the time of assessment. Time taken to achieve remission is reported.
Time Frame: Up to 12 months
Population: Efficacy analysis population. Number of participants analyzed = number of participants evaluable for this outcome.
Measure: Mean (Full Range); unit: days
Arm/Group | RA Cohort (Prospective)
Number analyzed (Participants) | 43
days | 130.31 [28 to 252]

8. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology (ACR) 20, ACR50, ACR70 and ACR90 Responses at Every Visit
Description: ACR20/ACR50/ACR70/ACR 90 response: greater than or equal to (≥) 20%/50%/70%/90% improvement in tender and swollen joint counts and 20%/50%/70%/90% improvement in 3 of the following 5 criteria: 1) Physician's global assessment of disease activity, 2) Participant assessment of disease activity, 3) Participant assessment of pain (VAS), 4) participant assessment of functional disability via a Health Assessment Questionnaire (HAQ), and 5) ESR at each visit.
Time Frame: Visit 3 (Week 4), Visit 4 (Week 8), Visit 5 (Week 12), Visit 6 (Week 16), Visit 7 (Week 20), Visit 8 (Week 24), Visit 9 (Week 28), Visit 10 (Week 32), Visit 11 (Week 36), Visit 12 (Week 42), Visit 13 (Week 44)
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | RA Cohort (Prospective)
Number analyzed (Participants) | 33
percentage of participants
  Visit 3: ACR 20 response (n=29) | 86.3
  Visit 3: ACR 50 response (n=29) | 10.3
  Visit 3: ACR 70 response (n=29) | 0
  Visit 3: ACR 90 response (n=29) | 0
  Visit 4: ACR 20 response (n=33) | 75.8
  Visit 4: ACR 50 response (n=33) | 18.2
  Visit 4: ACR 70 response (n=33) | 3.0
  Visit 4: ACR 90 response (n=33) | 0
  Visit 5: ACR 20 response (n=28) | 53.6
  Visit 5: ACR 50 response (n=28) | 28.6
  Visit 5: ACR 70 response (n=28) | 14.2
  Visit 5: ACR 90 response (n=28) | 0
  Visit 6: ACR 20 response (n=31) | 41.9
  Visit 6: ACR 50 response (n=31) | 35.5
  Visit 6: ACR 70 response (n=31) | 22.6
  Visit 6: ACR 90 response (n=31) | 0
  Visit 7: ACR 20 response (n=30) | 36.7
  Visit 7: ACR 50 response (n=30) | 26.7
  Visit 7: ACR 70 response (n=30) | 30.0
  Visit 7: ACR 90 response (n=30) | 0
  Visit 8: ACR 20 response (n=17) | 52.9
  Visit 8: ACR 50 response (n=17) | 23.5
  Visit 8: ACR 70 response (n=17) | 17.7
  Visit 8: ACR 90 response (n=17) | 0
  Visit 9: ACR 20 response (n=16) | 18.7
  Visit 9: ACR 50 response (n=16) | 56.3
  Visit 9: ACR 70 response (n=16) | 25.0
  Visit 9: ACR 90 response (n=16) | 0
  Visit 10: ACR 20 response (n=12) | 33.4
  Visit 10: ACR 50 response (n=12) | 33.3
  Visit 10: ACR 70 response (n=12) | 33.3
  Visit 10: ACR 90 response (n=12) | 0
  Visit 11: ACR 20 response (n=17) | 29.4
  Visit 11: ACR 50 response (n=17) | 23.5
  Visit 11: ACR 70 response (n=17) | 47.1
  Visit 11: ACR 90 response (n=17) | 0
  Visit 12: ACR 20 response (n=15) | 13.3
  Visit 12: ACR 50 response (n=15) | 46.7
  Visit 12: ACR 70 response (n=15) | 40.0
  Visit 12: ACR 90 response (n=15) | 0
  Visit 13: ACR 20 response (n=11) | 9.1
  Visit 13: ACR 50 response (n=11) | 27.3
  Visit 13: ACR 70 response (n=11) | 63.6
  Visit 13: ACR 90 response (n=11) | 0

9. Secondary Outcome: Change From Baseline (CFB) in ESR Values at Every Visit
Time Frame: Visit 2 (Baseline), Visit 3 (Week 4), Visit 4 (Week 8), Visit 5 (Week 12), Visit 6 (Week 16), Visit 7 (Week 20), Visit 8 (Week 24), Visit 9 (Week 28), Visit 10 (Week 32), Visit 11 (Week 36), Visit 12 (Week 40), Visit 13 (Week 44)
Population: Efficacy analysis population. Number of participants analyzed = number of participants evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: mm/hour
Arm/Group | RA Cohort (Prospective)
Number analyzed (Participants) | 27
mm/hour
  CFB at Visit 3 | -34.03 (30.87)
  CFB at Visit 4 | -39.63 (31.40)
  CFB at Visit 5 | -38.03 (32.07)
  CFB at Visit 6 | -38.71 (30.26)
  CFB at Visit 7 | -41.66 (33.23)
  CFB at Visit 8 | -39.07 (34.08)
  CFB at Visit 9 | -33.26 (37.61)
  CFB at Visit 10 | -35.89 (35.81)
  CFB at Visit 11 | -37.52 (32.42)
  CFB at Visit 12 | -40.37 (35.38)
  CFB at Visit 13 | -38.70 (35.32)
Statistical Analysis 1: Comparison: RA Cohort (Prospective); Statistical analysis for CFB at Visit 3; Test type: Superiority or Other; p = 0.001, Paired t-test
Statistical Analysis 2: Comparison: RA Cohort (Prospective); Statistical analysis for CFB at Visit 4; Test type: Superiority or Other; p = 0.001, Paired t-test
Statistical Analysis 3: Comparison: RA Cohort (Prospective); Statistical analysis for CFB at Visit 5; Test type: Superiority or Other; p = 0.001, Paired t-test
Statistical Analysis 4: Comparison: RA Cohort (Prospective); Statistical analysis for CFB at Visit 6; Test type: Superiority or Other; p = 0.001, Paired t-test
Statistical Analysis 5: Comparison: RA Cohort (Prospective); Statistical analysis for CFB at Visit 7; Test type: Superiority or Other; p = 0.001, Paired t-test
Statistical Analysis 6: Comparison: RA Cohort (Prospective); Statistical analysis for CFB at Visit 8; Test type: Superiority or Other; p = 0.001, Paired t-test
Statistical Analysis 7: Comparison: RA Cohort (Prospective); Statistical analysis for CFB at Visit 9; Test type: Superiority or Other; p = 0.001, Paired t-test
Statistical Analysis 8: Comparison: RA Cohort (Prospective); Statistical analysis for CFB at Visit 10; Test type: Superiority or Other; p = 0.001, Paired t-test
Statistical Analysis 9: Comparison: RA Cohort (Prospective); Statistical analysis for CFB at Visit 11; Test type: Superiority or Other; p = 0.001, Paired t-test
Statistical Analysis 10: Comparison: RA Cohort (Prospective); Statistical analysis for CFB at Visit 12; Test type: Superiority or Other; p = 0.001, Paired t-test
Statistical Analysis 11: Comparison: RA Cohort (Prospective); Statistical analysis for CFB at Visit 13; Test type: Superiority or Other; p = 0.001, Paired t-test

10. Secondary Outcome: Change From Baseline in C-Reactive Protein (CRP) Levels at Every Visit
Time Frame: as for outcome 9
Population: Efficacy analysis population. Number of participants analyzed = number of participants evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)
Arm/Group | RA Cohort (Prospective)
Number analyzed (Participants) | 17
milligrams per deciliter (mg/dL)
  CFB at Visit 3 | -12.34 (14.48)
  CFB at Visit 4 | -12.82 (16.24)
  CFB at Visit 5 | -13.77 (15.26)
  CFB at Visit 6 | -12.15 (18.24)
  CFB at Visit 7 | -16.51 (15.57)
  CFB at Visit 8 | -13.92 (18.98)
  CFB at Visit 9 | -12.79 (19.17)
  CFB at Visit 10 | -13.24 (18.53)
  CFB at Visit 11 | -14.74 (14.70)
  CFB at Visit 12 | -16.65 (15.17)
  CFB at Visit 13 | -15.69 (14.97)
Statistical Analysis 1: Comparison: RA Cohort (Prospective); Statistical analysis for CFB at Visit 3; Test type: Superiority or Other; p = 0.003, Paired t-test
Statistical Analysis 2: Comparison: RA Cohort (Prospective); Statistical analysis for CFB at Visit 4; Test type: Superiority or Other; p = 0.005, Paired t-test
Statistical Analysis 3: Comparison: RA Cohort (Prospective); Statistical analysis for CFB at Visit 5; Test type: Superiority or Other; p = 0.002, Paired t-test
Statistical Analysis 4: Comparison: RA Cohort (Prospective); Statistical analysis for CFB at Visit 6; Test type: Superiority or Other; p = 0.014, Paired t-test
Statistical Analysis 5: Comparison: RA Cohort (Prospective); Statistical analysis for CFB at Visit 7; Test type: Superiority or Other; p = 0.001, Paired t-test
Statistical Analysis 6: Comparison: RA Cohort (Prospective); Statistical analysis for CFB at Visit 8; Test type: Superiority or Other; p = 0.008, Paired t-test
Statistical Analysis 7: Comparison: RA Cohort (Prospective); Statistical analysis for CFB at Visit 9; Test type: Superiority or Other; p = 0.014, Paired t-test
Statistical Analysis 8: Comparison: RA Cohort (Prospective); Statistical analysis for CFB at Visit 10; Test type: Superiority or Other; p = 0.009, Paired t-test
Statistical Analysis 9: Comparison: RA Cohort (Prospective); Statistical analysis for CFB at Visit 11; Test type: Superiority or Other; p = 0.001, Paired t-test
Statistical Analysis 10: Comparison: RA Cohort (Prospective); Statistical analysis for CFB at Visit 12; Test type: Superiority or Other; p = 0.001, Paired t-test
Statistical Analysis 11: Comparison: RA Cohort (Prospective); Statistical analysis for CFB at Visit 13; Test type: Superiority or Other; p = 0.001, Paired t-test

11. Secondary Outcome: Participant's Global Assessment of Disease Activity Using VAS: Mean Change From Baseline at Every Visit
Description: The participant's global assessment of disease activity is assessed on a 0 to 100 mm horizontal VAS by the participant. The left-hand extreme of the line equals 0 mm, and is described as "no disease activity" (symptom-free and no arthritis symptoms) and the right-hand extreme equals 100 mm, and is described as "maximum disease activity" (maximum arthritis disease activity). A negative change from baseline indicated improvement.
Time Frame: as for outcome 9
Population: Efficacy analysis population. Number of participants analyzed = number of participants evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | RA Cohort (Prospective)
Number analyzed (Participants) | 41
millimeters
  CFB at Visit 3 | -11.34 (21.97)
  CFB at Visit 4 | -18.67 (26.29)
  CFB at Visit 5 | -17.86 (33.62)
  CFB at Visit 6 | -24.51 (35.40)
  CFB at Visit 7 | -25.90 (36.66)
  CFB at Visit 8 | -27.20 (37.13)
  CFB at Visit 9 | -28.17 (37.50)
  CFB at Visit 10 | -27.25 (37.07)
  CFB at Visit 11 | -30.71 (39.16)
  CFB at Visit 12 | -30.42 (38.13)
  CFB at Visit 13 | -30.34 (37.86)
Statistical Analysis 1: Comparison: RA Cohort (Prospective); Statistical analysis for CFB at Visit 3; Test type: Superiority or Other; p = 0.002, Wilcoxon sign rank test
Statistical Analysis 2: Comparison: RA Cohort (Prospective); Statistical analysis for CFB at Visit 4; Test type: Superiority or Other; p = 0.001, Wilcoxon sign rank test
Statistical Analysis 3: Comparison: RA Cohort (Prospective); Statistical analysis for CFB at Visit 5; Test type: Superiority or Other; p = 0.002, Wilcoxon sign rank test
Statistical Analysis 4: Comparison: RA Cohort (Prospective); Statistical analysis for CFB at Visit 6; Test type: Superiority or Other; p = 0.001, Wilcoxon sign rank test
Statistical Analysis 5: Comparison: RA Cohort (Prospective); Statistical analysis for CFB at Visit 7; Test type: Superiority or Other; p = 0.001, Wilcoxon sign rank test
Statistical Analysis 6: Comparison: RA Cohort (Prospective); Statistical analysis for CFB at Visit 8; Test type: Superiority or Other; p = 0.001, Wilcoxon sign rank test
Statistical Analysis 7: Comparison: RA Cohort (Prospective); Statistical analysis for CFB at Visit 9; Test type: Superiority or Other; p = 0.001, Wilcoxon sign rank test
Statistical Analysis 8: Comparison: RA Cohort (Prospective); Statistical analysis for CFB at Visit 10; Test type: Superiority or Other; p = 0.001, Wilcoxon sign rank test
Statistical Analysis 9: Comparison: RA Cohort (Prospective); Statistical analysis for CFB at Visit 11; Test type: Superiority or Other; p = 0.001, Wilcoxon sign rank test
Statistical Analysis 10: Comparison: RA Cohort (Prospective); Statistical analysis for CFB at Visit 12; Test type: Superiority or Other; p = 0.001, Wilcoxon sign rank test
Statistical Analysis 11: Comparison: RA Cohort (Prospective); Statistical analysis for CFB at Visit 13; Test type: Superiority or Other; p = 0.001, Wilcoxon sign rank test

12. Secondary Outcome: Physician's Global Assessment of Disease Activity Using VAS: Mean Change From Baseline at Every Visit
Description: The physician's global assessment of disease activity is assessed on a 0 to 100 mm horizontal VAS by the physician. The left-hand extreme of the line equals 0 mm, and is described as "no disease activity" (symptom-free and no arthritis symptoms) and the right-hand extreme equals 100 mm, and is described as "maximum disease activity" (maximum arthritis disease activity).
Time Frame: as for outcome 9
Population: Efficacy analysis population. Number of participants analyzed = number of participants evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | RA Cohort (Prospective)
Number analyzed (Participants) | 41
millimeters
  CFB at Visit 3 | -17.78 (19.72)
  CFB at Visit 4 | -23.56 (24.64)
  CFB at Visit 5 | -23.85 (33.00)
  CFB at Visit 6 | -29.06 (33.91)
  CFB at Visit 7 | -27.22 (34.90)
  CFB at Visit 8 | -29.00 (35.51)
  CFB at Visit 9 | -29.86 (36.32)
  CFB at Visit 10 | -28.68 (35.95)
  CFB at Visit 11 | -32.51 (37.57)
  CFB at Visit 12 | -32.10 (36.58)
  CFB at Visit 13 | -32.64 (36.93)
Statistical Analysis 1: Comparison: RA Cohort (Prospective); Statistical analysis for CFB at Visit 3; Test type: Superiority or Other; p = 0.001, Wilcoxon sign rank test
Statistical Analysis 2: Comparison: RA Cohort (Prospective); Statistical analysis for CFB at Visit 4; Test type: Superiority or Other; p = 0.001, Wilcoxon sign rank test
Statistical Analysis 3: Comparison: RA Cohort (Prospective); Statistical analysis for CFB at Visit 5; Test type: Superiority or Other; p = 0.001, Wilcoxon sign rank test
Statistical Analysis 4: Comparison: RA Cohort (Prospective); Statistical analysis for CFB at Visit 6; Test type: Superiority or Other; p = 0.001, Wilcoxon sign rank test
Statistical Analysis 5: Comparison: RA Cohort (Prospective); Statistical analysis for CFB at Visit 7; Test type: Superiority or Other; p = 0.001, Wilcoxon sign rank test
Statistical Analysis 6: Comparison: RA Cohort (Prospective); Statistical analysis for CFB at Visit 8; Test type: Superiority or Other; p = 0.001, Wilcoxon sign rank test
Statistical Analysis 7: Comparison: RA Cohort (Prospective); Statistical analysis for CFB at Visit 9; Test type: Superiority or Other; p = 0.001, Wilcoxon sign rank test
Statistical Analysis 8: Comparison: RA Cohort (Prospective); Statistical analysis for CFB at Visit 10; Test type: Superiority or Other; p = 0.001, Wilcoxon sign rank test
Statistical Analysis 9: Comparison: RA Cohort (Prospective); Statistical analysis for CFB at Visit 11; Test type: Superiority or Other; p = 0.001, Wilcoxon sign rank test
Statistical Analysis 10: Comparison: RA Cohort (Prospective); Statistical analysis for CFB at Visit 12; Test type: Superiority or Other; p = 0.001, Wilcoxon sign rank test
Statistical Analysis 11: Comparison: RA Cohort (Prospective); Statistical analysis for CFB at Visit 13; Test type: Superiority or Other; p = 0.001, Wilcoxon sign rank test

13. Secondary Outcome: Participant's Assessment of Pain Using VAS: Mean Change From Baseline at Every Visit
Description: The participant assessed their pain on a 0 to 100 mm horizontal VAS. The left-hand extreme of the line equals 0 mm, and is described as "no pain" and the right-hand extreme equals 100 mm, and is described as "unbearable pain". A negative change indicated improvement.
Time Frame: as for outcome 9
Population: Efficacy analysis population. Number of participants analyzed = number of participants evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | RA Cohort (Prospective)
Number analyzed (Participants) | 35
millimeters
  CFB at Visit 3 | -13.66 (19.43)
  CFB at Visit 4 | -20.93 (22.23)
  CFB at Visit 5 | -21.14 (26.46)
  CFB at Visit 6 | -26.34 (27.32)
  CFB at Visit 7 | -29.32 (27.19)
  CFB at Visit 8 | -29.75 (27.97)
  CFB at Visit 9 | -31.10 (28.21)
  CFB at Visit 10 | -30.17 (27.83)
  CFB at Visit 11 | -33.88 (30.19)
  CFB at Visit 12 | -33.71 (28.25)
  CFB at Visit 13 | -33.63 (28.33)
Statistical Analysis 1: Comparison: RA Cohort (Prospective); Statistical analysis for CFB at Visit 3; Test type: Superiority or Other; p = 0.001, Wilcoxon sign rank test
Statistical Analysis 2: Comparison: RA Cohort (Prospective); Statistical analysis for CFB at Visit 4; Test type: Superiority or Other; p = 0.001, Wilcoxon sign rank test
Statistical Analysis 3: Comparison: RA Cohort (Prospective); Statistical analysis for CFB at Visit 5; Test type: Superiority or Other; p = 0.001, Wilcoxon sign rank test
Statistical Analysis 4: Comparison: RA Cohort (Prospective); Statistical analysis for CFB at Visit 6; Test type: Superiority or Other; p = 0.001, Wilcoxon sign rank test
Statistical Analysis 5: Comparison: RA Cohort (Prospective); Statistical analysis for CFB at Visit 7; Test type: Superiority or Other; p = 0.001, Wilcoxon sign rank test
Statistical Analysis 6: Comparison: RA Cohort (Prospective); Statistical analysis for CFB at Visit 8; Test type: Superiority or Other; p = 0.001, Wilcoxon sign rank test
Statistical Analysis 7: Comparison: RA Cohort (Prospective); Statistical analysis for CFB at Visit 9; Test type: Superiority or Other; p = 0.001, Wilcoxon sign rank test
Statistical Analysis 8: Comparison: RA Cohort (Prospective); Statistical analysis for CFB at Visit 10; Test type: Superiority or Other; p = 0.001, Wilcoxon sign rank test
Statistical Analysis 9: Comparison: RA Cohort (Prospective); Statistical analysis for CFB at Visit 11; Test type: Superiority or Other; p = 0.001, Wilcoxon sign rank test
Statistical Analysis 10: Comparison: RA Cohort (Prospective); Statistical analysis for CFB at Visit 12; Test type: Superiority or Other; p = 0.001, Wilcoxon sign rank test
Statistical Analysis 11: Comparison: RA Cohort (Prospective); Statistical analysis for CFB at Visit 13; Test type: Superiority or Other; p = 0.001, Wilcoxon sign rank test

14. Secondary Outcome: Health Assessment Questionnaire Disability Index (HAQ-DI): Mean Change From Baseline at Every Visit
Description: HAQ-DI is a self-completed patient questionnaire specific for rheumatoid arthritis. It consists of 20 questions referring to 8 domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and common daily activities. Each domain has at least 2 component questions. There are 4 possible responses for each component 0=without any difficulty, 1=with some difficulty, 2=with much difficulty and 3=unable to do. The HAQ-DI is the sum of the scores from all domains and ranged from 0 (best) to 24 (worst). A negative change from baseline indicated improvement.
Time Frame: as for outcome 9
Population: Efficacy analysis population. Number of participants analyzed = number of participants evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | RA Cohort (Prospective)
Number analyzed (Participants) | 35
units on scale
  CFB at Visit 3 | -02.40 (09.08)
  CFB at Visit 4 | -02.21 (10.20)
  CFB at Visit 5 | -03.79 (13.43)
  CFB at Visit 6 | -03.85 (12.94)
  CFB at Visit 7 | -04.05 (10.67)
  CFB at Visit 8 | -03.92 (11.16)
  CFB at Visit 9 | -03.90 (11.68)
  CFB at Visit 10 | -03.11 (10.76)
  CFB at Visit 11 | -04.28 (12.40)
  CFB at Visit 12 | -04.35 (12.38)
  CFB at Visit 13 | -04.39 (12.37)
Statistical Analysis 1: Comparison: RA Cohort (Prospective); Statistical analysis for CFB at Visit 3; Test type: Superiority or Other; p = 0.064, Wilcoxon sign rank test
Statistical Analysis 2: Comparison: RA Cohort (Prospective); Statistical analysis for CFB at Visit 4; Test type: Superiority or Other; p = 0.104, Wilcoxon sign rank test
Statistical Analysis 3: Comparison: RA Cohort (Prospective); Statistical analysis for CFB at Visit 5; Test type: Superiority or Other; p = 0.052, Wilcoxon sign rank test
Statistical Analysis 4: Comparison: RA Cohort (Prospective); Statistical analysis for CFB at Visit 6; Test type: Superiority or Other; p = 0.043, Wilcoxon sign rank test
Statistical Analysis 5: Comparison: RA Cohort (Prospective); Statistical analysis for CFB of Visit 7; Test type: Superiority or Other; p = 0.015, Wilcoxon sign rank test
Statistical Analysis 6: Comparison: RA Cohort (Prospective); Statistical analysis for CFB at Visit 8; Test type: Superiority or Other; p = 0.023, Wilcoxon sign rank test
Statistical Analysis 7: Comparison: RA Cohort (Prospective); Statistical analysis for CFB at Visit 9; Test type: Superiority or Other; p = 0.028, Wilcoxon sign rank test
Statistical Analysis 8: Comparison: RA Cohort (Prospective); Statistical analysis for CFB at Visit 10; Test type: Superiority or Other; p = 0.048, Wilcoxon sign rank test
Statistical Analysis 9: Comparison: RA Cohort (Prospective); Statistical analysis for CFB at Visit 11; Test type: Superiority or Other; p = 0.025, Wilcoxon sign rank test
Statistical Analysis 10: Comparison: RA Cohort (Prospective); Statistical analysis for CFB at Visit 12; Test type: Superiority or Other; p = 0.023, Wilcoxon sign rank test
Statistical Analysis 11: Comparison: RA Cohort (Prospective); Statistical analysis for CFB at Visit 13; Test type: Superiority or Other; p = 0.022, Wilcoxon sign rank test

ADVERSE EVENTS:
Time Frame: Up to 12 months
Arm/Group | RA Cohort (Prospective + Retrospective)
Serious Adverse Events (participants affected / at risk) | 8/110
Other Adverse Events (participants affected / at risk) | 35/110
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RA Cohort (Prospective + Retrospective) (N=110)
Supraventricular Tachycardia (Cardiac disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Acute Gastroenteritis (Infections and infestations) | 1
Tuberculosis of Vertebral Column (Infections and infestations) | 1
Tibia Fracture (Injury, poisoning and procedural complications) | 1
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 1
Hip Arthroplasty (Injury, poisoning and procedural complications) | 1
Motor Peripheral Neuropathy (Nervous system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RA Cohort (Prospective + Retrospective) (N=110)
Leucopenia (Blood and lymphatic system disorders) | 6
Eosinophilia (Blood and lymphatic system disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Eye Inflammation (Eye disorders) | 1
Eye Swelling (Eye disorders) | 1
Fever (General disorders) | 2
General Body Pain (General disorders) | 1
Redness (General disorders) | 1
Swelling Face (General disorders) | 1
Rash (General disorders) | 4
Oedema Peripheral (Metabolism and nutrition disorders) | 1
Pain In Limb (Musculoskeletal and connective tissue disorders) | 1
Painful Joints (Musculoskeletal and connective tissue disorders) | 1
Fracture (Musculoskeletal and connective tissue disorders) | 1
Stiffness (Musculoskeletal and connective tissue disorders) | 1
Acute Gastroenteritis (Infections and infestations) | 2
Upper Respiratory Tract Infection (Infections and infestations) | 1
Application Site Pustules (Infections and infestations) | 1
Transaminitis (Investigations) | 1
Liver Enzyme Abnormal (Investigations) | 1
Lipids Increased (Investigations) | 1
Weight Gain (Investigations) | 1
Generalized Itching (Skin and subcutaneous tissue disorders) | 1
Itching (Skin and subcutaneous tissue disorders) | 5
Urticarial Rash (Skin and subcutaneous tissue disorders) | 2
Parasthesia (Nervous system disorders) | 1
Giddiness (Nervous system disorders) | 2
Insomnia (Nervous system disorders) | 1
Per Vaginal Bleeding (Reproductive system and breast disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.